CLINICAL TRIAL: NCT00642642
Title: A Phase II/III Double-Blind, Randomized, Placebo-Controlled Trial of the Safety and Efficacy of Isolagen Therapy in the Treatment of Moderate to Sever Facial Acne Scarring
Brief Title: Safety and Efficacy Study of Autologous Fibroblasts in the Treatment of Severe Facial Acne Scarring
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IT-A-008
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-07

CONDITIONS: Acne Scarring of the Face
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double blinded active (Experimental): Subject will receive autologous fibroblast treatment on either their left or right side of their face
  Interventions: Biological: Autologous Human Fibroblasts (azficel-T)
- Double blinded placebo (Placebo Comparator): Subject will receive placebo treatment on the opposite side of the face from active treatment
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Autologous Human Fibroblasts (azficel-T) — 1. Collection of 3 mm post auricular skin punch biopsies.
  2. Administration of 3 study treatments administered 14 ± 7 days apart.
  Other Names: LAVIV
  Arms: Double blinded active
Biological: Placebo — 1. Collection of 3 mm post auricular skin punch biopsies.
  2. Administration of 3 study treatments administered 14 ± 7 days apart.
  Arms: Double blinded placebo

SUMMARY:
The purpose of this study is to evaluate the safety profile and the treatment effect of Isolagen TherapyTM and placebo when administered to facial acne scars.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 years and 65 years of age.
2. Investigator assessment of the acne scarring on each cheek of moderate to severe.
3. A history of acne scarring for more than 3 years.
4. Subject assesses the appearance of both sides of their facial acne scars as dissatisfied or very dissatisfied with appearance.

Exclusion Criteria:

1. Significant active acne.
2. Use of oral antibiotic or retinoid active acne therapy within one year of enrollment.
3. Presence of hypertrophic scars on the cheeks.
4. More than 20% of treatment area comprised of ice pick scars or sinus tracts
5. Treatment area per cheek is less than 9 cm x cm
6. Unilateral or unbalanced acne scar distribution.
7. Physical attributes which prevent the assessment or treatment of the acne scars.
8. Treatment with an investigational product or procedure within 30 days prior to study enrollment or plans to participate in another clinical trial during the course of this study.
9. Previous treatment with Isolagen TherapyTM.
10. Use of Isotretinoin within one year of enrollment into study.
11. Use of permanent or semi-permanent dermal fillers in the treatment areas within defined time frames.
12. Disorders or drugs that increase bleeding or clotting.
13. Pregnant or lactating women or women trying to become pregnant during the study.
14. Excessive exposure to sun.
15. Smoking more than ½ pack of cigarettes per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Brighton Medical Corporation, Beverly Hills, California
  - Therapeutics Clinical Research, San Diego, California
  - The Laser Institute for Dermatology, Santa Monica, California
  - Dermatology Research Institute, LLC, Coral Gables, Florida
  - Maryland Laser, Skin and Vein Institute, Hunt Valley, Maryland
  - Sadick Dermatology, New York, New York
  - Dermatology, Laser and Vein Specialists of the Carolinas, Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 7 Nov 2007 and 6 March 2008
Pre-assignment Details: Patients were enrolled and biopsied for manufacture of study product. Patients for whom study product could not be manufactured were excluded from the Intent to Treat (ITT) population.
Groups:
- Autologous Fibroblasts and Placebo: Patients were treated with autologous fibroblasts on one cheek, and placebo on the opposite cheek
Period: Biopsy & Product Manufacture
Arm/Group | Autologous Fibroblasts and Placebo
Started | 122
Completed | 109 (Patients biopsied and for whom study product could be produced are considered completed)
Not Completed | 13
Period: Treatment & Follow Up
Arm/Group | Autologous Fibroblasts and Placebo
Started | 109
Completed | 92
Not Completed | 17
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Fibroblasts and Placebo
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 109
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.7 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 78
  More than one race | 0
  Unknown or Not Reported | 17

OUTCOME MEASURES:

1. Primary Outcome: Evaluator Live Acne Scarring Assessment Responders
Description: Subjects who improved by 1 point or more on the Evaluator Live Acne Scarring Assessment (ELASA), as assessed by the evaluating Investigator, are counted as responders. On the ELASA scale, a score of 0 (Clear) is best and a score of 4 (Severe) is worst.
Time Frame: Baseline (prior to first treatment) and four months after last treatment
Population: Analysis population was the ITT population, defined as subjects for whom product could be produced and who were randomized to study treatment, whether or not all study treatments are actually received.
Measure: Number; unit: Participants
Groups:
- Autologous Fibroblasts Cheeks: Cheeks treated with autologous fibroblasts (azficel-T)
- Placebo Cheeks: Cheeks treated with placebo solution
Arm/Group | Autologous Fibroblasts Cheeks | Placebo Cheeks
Number analyzed (Participants) | 109 | 109
Participants | 64 | 46
Statistical Analysis 1: Comparison: Autologous Fibroblasts Cheeks vs Placebo Cheeks; Null hypothesis: no difference in the response rates between the two treatment arms. Statistical test: McNemar's paired test of proportions Significance level: two sided alpha of 0.05 for each of the two co-primary endpoints. Assumptions for power calculations: Response rate for azficel-T treated cheek = 40% Response rate for placebo treated cheek = 20% 10% dropout rate; dropouts counted as failures. Low correlation between cheeks & 50% correlation between endpoints; Test type: Superiority or Other; p = 0.0109, McNemar — a priori threshold for statistical significance was 0.05; Paired test of proportions

2. Primary Outcome: Subject Live Acne Scarring Assessment Responders
Description: Cheeks that improved by at least two points on the Subject Live Acne Scarring Assessment (SLASA) as scored by the subject were considered responders. On the SLASA scale, a score of -2 (Very Dissatisfied) was worst and a score of 2 (Very Satisfied) was best.
Time Frame: Baseline (prior to first treatment) and four months after last treatment
Population: Analysis was performed on the ITT population
Measure: Number; unit: Cheeks
Groups:
- Autologous Fibroblast Cheeks: Cheeks treated with autologous fibroblasts
Arm/Group | Autologous Fibroblast Cheeks | Placebo Cheeks
Number analyzed (Participants) | 109 | 109
Cheeks | 47 | 20
Statistical Analysis 1: Comparison: Autologous Fibroblast Cheeks vs Placebo Cheeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, McNemar — a priori threshold for statistical significance = 0.05; paired test of proportions

3. Secondary Outcome: Evaluator Live Acne Scarring Assessment Responders
Description: as for outcome 1
Time Frame: Baseline (prior to first treatment) compared to one, two, and three months after last treatment
Population: Number of cheeks for analysis was the ITT population
Measure: Number; unit: Participants
Arm/Group | Autologous Fibroblasts Cheeks | Placebo Cheeks
Number analyzed (Participants) | 109 | 109
Participants
  1 Month Post Treatment | 54 | 32
  2 Months Post Treatment | 56 | 41
  3 Months Post Treatment | 57 | 47

4. Secondary Outcome: Subject Live Acne Scarring Assessment Responders
Description: as for outcome 2
Time Frame: Baseline (prior to first treatment) compared to one, two, and three months after last treatment
Population: Analysis was performed on the ITT population
Measure: Number; unit: Cheeks
Groups:
- Autologous Fibroblast Cheeks: Cheeks randomized to receive autologous fibroblast treatment
- Placebo Cheeks: Cheeks randomized to receive placebo treatment
Arm/Group | Autologous Fibroblast Cheeks | Placebo Cheeks
Number analyzed (Participants) | 109 | 109
Cheeks
  1 Month Post Treatment | 34 | 10
  2 Months Post Treatment | 41 | 15
  3 Months Post Treatment | 43 | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of patient biopsy through the final study visit, four months after final study treatment (five months after first study treatment).
Groups:
- Non-treatment Area Adverse Events: Systemic adverse events and adverse events that occured outside of the study treatment area will be reported in this group
Arm/Group | Autologous Fibroblast Cheeks | Placebo Cheeks | Non-treatment Area Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/122 | 1/122
Other Adverse Events (participants affected / at risk) | 11/122 | 10/122 | 1/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Fibroblast Cheeks (N=122) | Placebo Cheeks (N=122) | Non-treatment Area Adverse Events (N=122)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Patient treated for overdose of recreational drugs after being biopsied and enrolled in the study, but prior to receiving any study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Fibroblast Cheeks (N=122) | Placebo Cheeks (N=122) | Non-treatment Area Adverse Events (N=122)
Erythema (Skin and subcutaneous tissue disorders) | 11 (33) | 10 (29) | 1 (1) — Administration site condition
Swelling (General disorders) | 10 (29) | 10 (29) | 1 (1) — Administration site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications or presentations by the Investigator or his associates, were required to be submitted to the sponsor for review and approval prior to publication or presentation in any form.